CLINICAL TRIAL: NCT05105581
Title: Psychiatric Comorbidity and Quality of Life in Patients With Obsessive Compulsive Disorder(Case Control Study )
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Safwat AbdElrhman, Assistant Professor of Psychiatry, Assiut University
Other Study IDs: Assiut Unirvesity Hospital
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Patients): Patients: 37 patients with OCD diagnosed according to DSM-5
  1. Inclusion criteria:
     1. both sex
     2. age groups : 18 : 60 are included
     3. accept to participate in the study
  2. Exclusion criteria
     1. presence of major neurological disease as head trauma and sensory or motor defect as blindness or deafness
     2. Active psychiatric disordes
     3. patients refuse to participate in the study
- Group 2 (Controlled): 37 healthy populations matched with PT group in age , sex , socioeconomic state
  Interventions: Behavioral: Quality of life scale

INTERVENTIONS:
Behavioral: Quality of life scale — 1. To assess the quality of life of patient
  2. To assess the degree of OCD
  Other Names: Yale-Brown Obsessive-Compulsive Scale
  Groups: Group 2 (Controlled)

SUMMARY:
Psychiatric Comorbidity and quality of life in patients with Obsessive Compulsive Disorder(case control study )

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a mental and behavioral disorder[7] in which a person has certain thoughts repeatedly (called "obsessions") and/or feels the need to perform certain routines repeatedly (called "compulsions") to an extent that generates distress or impairs general functioning.[1][2] The person is unable to control either the thoughts or activities for more than a short period of time.[1] Common compulsions include excessive hand washing, the counting of things, and checking to see if a door is locked.[1] These activities occur to such a degree that the person's daily life is negatively affected,[1] often taking up more than an hour a day.[2] Most adults realize that the behaviors do not make sense.[1] The condition is associated with tics, anxiety disorder, and an increased risk of suicide.[2][3] The cause is unknown.[1] There appear to be some genetic components, with both identical twins more often affected than both non-identical twins.[2] Risk factors include a history of child abuse or other stress-inducing event.[2] Some cases have been documented to occur following infections.[2] The diagnosis is based on the symptoms and requires ruling out other drug-related or medical causes.[2] Rating scales such as the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) can be used to assess the severity.[8] Other disorders with similar symptoms include anxiety disorder, major depressive disorder, eating disorders, tic disorders, and obsessive-compulsive personality disorder.[2]

Treatment may involve psychotherapy, such as cognitive behavioral therapy (CBT), and antidepressants, such as selective serotonin reuptake inhibitors (SSRIs) or clomipramine.[4][5] CBT for OCD involves increasing exposure to fears and obsessions while preventing the compulsive behavior that would normally accompany the obsessions.[4] Contrary to this, metacognitive therapy encourages the ritual behaviors in order to alter the relationship to one's thoughts about them.[9] While clomipramine appears to work as well as do SSRIs, it has greater side effects and thus is typically reserved as a second-line treatment.[4] Atypical antipsychotics may be useful when used in addition to an SSRI in treatment-resistant cases but are also associated with an increased risk of side effects.[5][10] Without treatment, the condition often lasts decades.[2]

ELIGIBILITY:
Inclusion Criteria:

* 1. both sex 2. age groups : 18 : 60 are included 3. accept to participate in the study

Exclusion Criteria:

- 1. presence of major neurological disease as head trauma and sensory or motor defect as blindness or deafness

2. Active psychiatric disordes 3. patients refuse to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Psychiatric interview
  2. Diagnosis : according to DSM-.5 using Yale-Brown Obsessive-Compulsive Scale for diagnosis and severity
  3. Psychiatric comorbidity :
     SCID I -SCID II scale
  4. Socioeconomic state
  5. Quality of life scale
  6. EEG
Sampling Method: Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
quality of life scale | about 6 months
  assess the quality of life in OCD patients

IPD SHARING:
Plan to Share IPD: No